CLINICAL TRIAL: NCT04915235
Title: Prevalence and Prognosis of Cardiac Amiloidosis in Turkey- Registry Study
Brief Title: Prevalence and Prognosis of Cardiac Amiloidosis in Turkey
Acronym: PAPCAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turkish Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: PAPCAT
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial | interventions — Algorithms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Algorithm — Algorithm

SUMMARY:
Patients with left ventricular hypertrophy are further examined according to an algorithm to check if they have a cardiac amyloidosis

ELIGIBILITY:
Inclusion Criteria:

* Patients with left ventricular hypertrophy without left ventricular pressure or volume (IVS≥13mm)
* Patients with left ventricular hypertrophy and hypertension or aortic stenosis without left ventricular pressure or volume (IVS>15mm)

Exclusion Criteria:

* Patients with left ventricular pressure or volume except the ones with aortic stenosis and arterial hypertension
* Patients with sigmoid septum and their hypertrophy limited in sigmoid area
* Patients with highly probable sarcometric hypertrophy cardiomyopathy confirmed with LV morhpology and genetic testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left ventricular hypertrophy
Sampling Method: Probability Sample
Enrollment: 2087 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Amyloidosis | Upon screening
  Patients with left ventricular hypertrophy and Cardiac Amyloidosis

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Faculty of Medicine, Izmir, Turkey (Türkiye)